CLINICAL TRIAL: NCT02308527
Title: A Randomised Phase IIb Trial of Bevacizumab Added to Temozolomide ± Irinotecan for Children With Refractory/Relapsed Neuroblastoma - BEACON-Neuroblastoma Trial
Brief Title: Activity Study of Bevacizumab With Temozolomide ± Irinotecan for Neuroblastoma in Children
Acronym: BEACON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry); Imagine for Margo (Unknown); EUSA Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RG_11-087; 2012-000072-42 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-12-04 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Neuroblastoma
Keywords: Children; Young adults
MeSH Terms: conditions — Neuroblastoma | interventions — Bevacizumab; Temozolomide; Irinotecan; Topotecan; dinutuximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Temozolomide (Active Comparator): Temozolomide Days 1-5 every 4 weeks
  Interventions: Drug: Temozolomide
- Bevacizumab + Temozolomide (Experimental): Bevacizumab Day 1 and 15 + Temozolomide Days 1-5 every 4 weeks
  Interventions: Drug: Bevacizumab; Drug: Temozolomide
- Irinotecan + Temozolomide (Experimental): Irinotecan Days 1-5 + Temozolomide Days 1-5 every 3 weeks
  Interventions: Drug: Temozolomide; Drug: Irinotecan
- Bevacizumab + Irinotecan + Temozolomide (Experimental): Bevacizumab Day 1 + Irinotecan Days 1-5 + Temozolomide Days 1-5 every 3 weeks
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Drug: Bevacizumab
- Temozolomide + Topotecan (Experimental): Temozolomide Days 1-5+ Topotecan Days 1-5 every 4 weeks
  Interventions: Drug: Topotecan; Drug: Temozolomide
- Bevacizumab + Temozolomide + Topotecan (Experimental): Bevacizumab Day 1 and 15 + Temozolomide Days 1-5 + Topotecan Days 1-5 every 4 weeks
  Interventions: Drug: Bevacizumab; Drug: Topotecan; Drug: Temozolomide
- Dinutuximab beta + Temozolomide (Experimental): Dinutuximab beta Days 1-7 + Temozolomide Days 1-5 every 4 weeks
  Interventions: Drug: Temozolomide; Drug: Dinutuximab Beta
- Dinutuximab beta + Temozolomide + Topotecan (Experimental): Dinutuximab beta Days 1-7 + Temozolomide Days 1-5 + Topotecan Days 1-5 every 4 weeks
  Interventions: Drug: Temozolomide; Drug: Topotecan; Drug: Dinutuximab Beta
- Dinutuximab beta + Topotecan + Cyclophosphamide (Other): Dinutuximab beta Days 1-7 + Topotecan Days 1-5 + Cyclophosphamide Days 1-5 every 4 weeks
  Interventions: Drug: Topotecan; Drug: Dinutuximab Beta; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bevacizumab — 10mg/kg IV (in the vein) on Days 1 and 15 of a 4 week cycle, for 6 cycles or until progression
  Other Names: Avastin
  Arms: Bevacizumab + Temozolomide; Bevacizumab + Temozolomide + Topotecan
Drug: Temozolomide — 200mg/m2/d PO (capsule taken orally) on Days 1 to 5 of a 4 week cycle, for 6 cycles or until progression
  Other Names: Temodal
  Arms: Bevacizumab + Temozolomide; Dinutuximab beta + Temozolomide; Dinutuximab beta + Temozolomide + Topotecan; Temozolomide
Drug: Temozolomide — 100mg/m2/d PO (capsule taken orally) on Days 1 to 5 of a 3 week cycle, for 6 cycles or until progression
  Other Names: Temodal
  Arms: Bevacizumab + Irinotecan + Temozolomide; Irinotecan + Temozolomide
Drug: Irinotecan — 50mg/m2/d IV (in the vein) on Days 1 to 5 of a 3 week cycle, for 6 cycles or until progression
  Other Names: Campto
  Arms: Bevacizumab + Irinotecan + Temozolomide; Irinotecan + Temozolomide
Drug: Bevacizumab — 15mg/kg IV (in the vein) on Day 1 of a 3 week cycle, for 6 cycles or until progression
  Other Names: Avastin
  Arms: Bevacizumab + Irinotecan + Temozolomide
Drug: Topotecan — 0.75mg/m2/d IV (in the vein) on Days 1-5 of a 4 week cycle, for 6 cycles or until progression
  Arms: Bevacizumab + Temozolomide + Topotecan; Dinutuximab beta + Temozolomide + Topotecan; Dinutuximab beta + Topotecan + Cyclophosphamide; Temozolomide + Topotecan
Drug: Temozolomide — 150mg/m2/d PO (capsule taken orally) on Days 1 to 5 of a 4 week cycle, for 6 cycles or until progression
  Other Names: Temodal
  Arms: Bevacizumab + Temozolomide + Topotecan; Temozolomide + Topotecan
Drug: Dinutuximab Beta — 10mg/m2/d IV (in the vein) on Days 1 to 7 of a 4 week cycle, for 6 cycles or until progression
  Other Names: Qarziba
  Arms: Dinutuximab beta + Temozolomide; Dinutuximab beta + Temozolomide + Topotecan; Dinutuximab beta + Topotecan + Cyclophosphamide
Drug: Cyclophosphamide — 250mg/m2/d IV (in the vein) on Days 1 to 5 of a 4 week cycle, for 6 cycles or until progression
  Arms: Dinutuximab beta + Topotecan + Cyclophosphamide

SUMMARY:
The purpose of this study is to investigate whether Bevacizumab (an anti-VEGF monoclonal antibody) added to a backbone chemotherapy regimen (Temozolomide, Irinotecan-Temozolomide or Topotecan-Temozolomide) demonstrates activity in children with relapsed or refractory neuroblastoma. Also, to investigate whether the addition of Irinotecan or Topotecan to Temozolomide increases the activity of chemotherapy.The primary objective of the study is the best response (Complete Response or Partial Response) while trial treatment, within 18 or 24 weeks depending on the arm of the trial the participant is randomised to. Secondary endpoints are assessing the side effects, the length of time before progression (Progression Free Survival) and overall survival (OS).

This trial will address two important questions:

* does targeting blood vessel development using bevacizumab, (a monoclonal antibody against the Vascular Endothelial Growth Factor (VEGF)), add to the effect on a tumour when used with existing chemotherapy, compared to the effect of the existing chemotherapy alone (temozolomide)? NOTE- This question has been completed.
* does the addition of a second chemotherapy drug (irinotecan or topotecan) increase the effect on a tumour compared to the effect of one alone (temozolomide) NOTE - This question has been completed.
* does the addition of dinutuximab beta added to a backbone chemotherapy (temozolomide or temozolomide + topotecan) increase the effect of backbone alone.

Patients aged 1-21 years of age with relapsed or refractory high-risk neuroblastoma are randomised to one of two treatment arms: temozolomide-topotecan (TTo) or dinutuximab beta-temozolomide-topotecan (dBTTo). Temozolomide (T), irinotecan-temozolomide (IT), bevacizumab-T (BT), BIT (bevacizumab-IT), bevacizumab-temozolomide-topotecan (BTTo) and dinutuximab beta-temozolomide (dBT) are now closed to recruitment.

DETAILED DESCRIPTION:
This is an international open-label, randomised, multicentre phase II trial of temozolomide ± irinotecan, with or without bevacizumab, for the treatment of patients with relapsed or refractory neuroblastoma. The study will evaluate the safety and activity of these combinations.

Patients will be registered into the trial and randomised at the same time to one of the following two arms (approximately 30 patients per arm):

TTo: Temozolomide + Topotecan dBTTo: Dinuximab beta + Temozolomide + Topotecan

Arms which have now closed to recruitment:

dBT: Dinutuximab beat + Temozolomide Closed 28 ]Jan 2020 T: Temozolomide - Closed 28 Jan 2020 BT: Bevacizumab + Temozolomide - Closed 7 Feb 2019 IT: Irinotecan + Temozolomide - Closed 21 June 2018 BIT: Bevacizumab + Irinotecan + Temozolomide - Closed 21 June 2018 BTTo: Bevacizumab + Temozolomide + Topotecan - Closed 7 Feb 2019

Randomisation will be via a secure on-line computer-based system at the Cancer Research Clinical Trial Unit (CRCTU), University of Birmingham, United Kingdom (UK) and patients will be allocated in a 2:1 ratio. Minimisation will be used to ensure balance across the arms for the important prognostic factors as described by London et al. [10]: a) relapsed, refractory disease, b) early (< 18 months), late relapse (≥18 months) and c) measurable versus evaluable disease (i.e. disease evaluated according to RECIST versus disease detectable only by MIBG scanning with or without bone marrow involvement as detected by local morphology) Patients will receive treatment for 6 courses, lasting 24 weeks.

Patients with a response (CR, PR) or stable disease (SD) while on the BEACON-Neuroblastoma trial will receive 6 cycles of trial treatment. If the patient has achieved a satisfactory response (i.e. CR, PR or SD) with acceptable toxicity, treatment may be extended beyond 6 cycles (up to 12 cycles) after discussion with the Sponsor and the Chief Investigator (CI).

In addition, patients randomised to TTo may recieve an optional regimen of dinutuximab beta + topotecan + cyclophosphamide (up to 6 cycles).

ELIGIBILITY:
Inclusion Criteria

* Histologically proven neuroblastoma as per International Neuroblastoma Staging System (INSS) definition
* Relapsed: any relapsed or progressed high-risk neuroblastoma
* Refractory high risk disease: Lack of adequate response to frontline therapy that precludes the patient from proceeding to consolidation therapies
* Measurable disease by cross sectional imaging (RECIST) or evaluable disease
* Age ≥1 to ≤21 years
* Informed consent from patient, parent or guardian
* Performance Status:Lansky ≥ 50%, Karnofsky ≥ 50% or Eastern Cooperative Oncology Group ≤3 (Patients who are unable to walk because of paralysis, but who are able to sit upright unassisted in a wheelchair, will be considered ambulatory for the purpose of assessing performance score)
* Life expectancy of ≥12 weeks
* No bone marrow disease: Platelets ≥75 x 10^9/L (unsupported for 72 hours), absolute neutrophil count ≥0.75 x10^9/L (no G-cerebrospinal fluid support for 72 hours), Haemoglobin ≥8 g/dL (transfusions allowed) Bone marrow disease: Platelets ≥50 x10^9/L (unsupported for 72 hours), absolute neutrophil count (ANC) ≥0.5 x 10^9/L (no granulocyte colony stimulating factor (G-CSF) for 72 hours), Haemoglobin ≥8 g/dL (transfusions allowed)
* Renal function (within 72 hours of eligibility assessment): Absence of clinically significant proteinuria (early morning urine dipstick <2+). When the dipstick urinalysis shows a proteinuria ≥2+, a protein:creatinine (Pr/Cr) ratio must be <0.5 or a 24 hour protein excretion must be <0.5g
* Serum creatinine ≤ 1.5 upper limit of normal for age, if higher, a calculated glomerular filtration rate (radioisotope) must be ≥60 ml/min/1.73 m2
* Liver function (within 72 hours of eligibility assessment): aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤2.5 ULN and Total bilirubin ≤1.5 upper limit of normal (ULN). In case of liver metastases, AST or ALT ≤5 ULN and Total bilirubin ≤2.5 ULN
* Cardiac function, shortening fraction ≥29% on echocardiogram
* Coagulation, patients not on anticoagulation must have an international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5 ULN for age. Anti-coagulation is permitted as long as the INR or APTT is within therapeutic limits (according to the medical standard of the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks at the time of study enrolment
* Blood pressure below 95th centile for age and sex. Use of antihypertensive medication is permitted
* Males or females of reproductive potential may not participate unless they agree to use an effective contraceptive method, for the duration of study therapy and for up to 6 months after the last dose of trial drugs. A negative urine pregnancy test must be obtained within 72 hours prior to dosing in females who are post-menarche
* No dyspnoea at rest and pulse oximetry > 94% in room air
* Availability and willingness to place a double central venous access if needed for trial treatment and supportive care in case of treatment with chemo-immunotherapy

Exclusion Criteria:

* Previous treatment with bevacizumab, temozolomide, irinotecan or any combination of these drugs
* Known hypersensitivity to: Any study drug or component of the formulation, Chinese hamster ovary products or other recombinant human or humanised antibodies, Dacarbazine
* Prior severe arterial thrombo-embolic events (e.g. cardiac ischemia, cerebral vascular accident, peripheral arterial thrombosis)
* Any ongoing arterial thrombo-embolic events
* Patient less than (at point of planned date of randomisation): 48 hours post bone marrow aspirate/trephine, 48 hours post central line insertion, Four weeks post major surgery, One week post core biopsy, Two weeks from prior chemotherapy, Six weeks from prior craniospinal radiotherapy or MIBG therapy and two weeks from radiotherapy to the tumour bed, Eight weeks from prior myeloablative therapy with haematopoietic stem cell rescue (autologous stem cell transplant), Three months from prior allogeneic stem cell transplant, 14 days or 5 half-lives (whichever occurs later) from last administration of an IMP in an IMP-trial, 6 months from presentation of lung haemorrhage/haemoptysis
* Bleeding metastases (patients with CNS metastases can be enrolled as long as the metastases are not bleeding)
* Invasion of major blood vessels
* Use of enzyme inducing anticonvulsants within 72 hours of randomisation
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation)
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding within 6 months prior to study enrolment
* Current chronic intestinal inflammatory disease/bowel obstruction
* Intolerance to galactose and fructose, lactase deficiency, and/or defect of absorption of galactose and fructose
* Pregnant or lactating patient
* Any uncontrolled medical condition that poses an additional risk to the patient (i.e. haemoptysis, non-healing, bone fracture, wound/ulcer)
* Low probability of treatment compliance
* Any uncontrolled medical condition that poses an additional risk to the patient
* Planned immunisation with live vaccine

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Best response (Complete Response or Partial Response) while on trial treatment, within 18 or 24 weeks depending on the arm of the trial participant is randomised to. | Within 18 or 24 weeks depending on the arm of the trial the participant is randomised to.
  To test whether bevacizumab added to a backbone chemotherapy regimen (temozolomide, irinotecan-temozolomide or topotecan-temozolomide) demonstrates activity in children with relapsed or refractory neuroblastoma To test whether the addition of irinotecan to temozolomide increases the activity of chemotherapy in children with relapsed or refractory neuroblastoma
For the bevacizumab part 2 only; Progression-free survival (PFS) | Assessment will be after 30 days after treatment or end of trial
  Progression-free survival (PFS)

SECONDARY OUTCOMES:
To evaluate the toxicity of the regimens | Assessment will be after 30 days after treatment or end of trial
  Safety of the regimens: Incidence and severity of Adverse Events (AE)s
To evaluate the safety of the regimens | Assessment will be after 30 days after treatment or end of trial
  Safety of the regimens: Progression-free survival (PFS)
To evaluate the overall safety of the regimens | Assessment will be after 30 days after treatment or end of trial
  Safety of the regimens: Overall survival (OS)
To evaluate the safety of the regimens | Assessment will be after 30 days after treatment or end of trial
  Safety of the regimens: Event-free survival (EFS)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Moreno, MD, Principal Investigator — University of Birmingham
Locations (10):
- St Anna Children's Hospital and CCRI/Studies and Statistics, Vienna, Austria
- University Hospital, Ghent, Belgium
- University Hospital Rigshospitalet, Copenhagen, Denmark
- Hopital des Enfants, Toulouse, France
- Our Ladys Children's Hospital Dublin, Dublin, Ireland
- Ospedale Pediatrico Bambino Gseu, Rome, Italy
- Natasha van Eijkelenburg, Utrecht, Netherlands
- Instituto de Investigacion Sanitaria, Valencia, Spain
- Swiss Paediatric Oncology Group, Bern, Switzerland
- The Royal Marsden NHS Foundation Trust and Institute of Cancer Research, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno L, Weston R, Owens C, Valteau-Couanet D, Gambart M, Castel V, Zwaan CM, Nysom K, Gerber N, Castellano A, Laureys G, Ladenstein R, Rossler J, Makin G, Murphy D, Morland B, Vaidya S, Thebaud E, van Eijkelenburg N, Tweddle DA, Barone G, Tandonnet J, Corradini N, Chastagner P, Paillard C, Bautista FJ, Gallego Melcon S, De Wilde B, Marshall L, Gray J, Burchill SA, Schleiermacher G, Chesler L, Peet A, Leach MO, McHugh K, Hayes R, Jerome N, Caron H, Laidler J, Fenwick N, Holt G, Moroz V, Kearns P, Gates S, Pearson ADJ, Wheatley K; Innovative Therapies for Children with Cancer (ITCC) and European Association for Neuroblastoma Research (SIOPEN). Bevacizumab, Irinotecan, or Topotecan Added to Temozolomide for Children With Relapsed and Refractory Neuroblastoma: Results of the ITCC-SIOPEN BEACON-Neuroblastoma Trial. J Clin Oncol. 2024 Apr 1;42(10):1135-1145. doi: 10.1200/JCO.23.00458. Epub 2024 Jan 8. PMID 38190578